CLINICAL TRIAL: NCT04863534
Title: Qualitative Muscular Ultrasound in covid19 ARDS Patients
Brief Title: Ultrasound Grayscale Analysis in ARDS covid19
Acronym: Graycovid
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Davide Chiumello, PROFESSOR, University of Milan
Other Study IDs: Umilan1
Record Dates: First submitted 2021-04-22; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Muscular Diseases; COVID-19 Acute Respiratory Distress Syndrome
Keywords: Ards; Covid 19; Muscular ultrasound
MeSH Terms: conditions — Muscular Diseases; Acute Lung Injury; COVID-19 | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasound — Muscular grayscale ultrasound

SUMMARY:
Recent evidence regarding the novel coronavirus disease 2019 (COVID19) is growing in describing the characteristics of this disease, with main focus on lung morphology. Few data are available regarding the peripheral and respiratory muscular characteristics. Using a ultrasound greyscale analysis, It Is possibile to evaluated the muscle quality.

The hypothesis of this studi is that a combined assessment of respiratory (i.e., intercostal and diaphragm) and peripheral (i.e., quadriceps) muscles quantity (as measured by thickness) and quality (as assessed by greyscale analysis), would reflect the severity of illness. Thus,the aims of this study are to assess if the quality characteristics of parasternal intercostal, diaphragm and quadriceps muscles of ICU COVID19 patients influenced the outcomes and are correlated with other variables, such as fluid or protein balance, or indexes of inflammation

DETAILED DESCRIPTION:
Up to 30% of the patients affected by the novel coronavirus disease 2019 (COVID19) may develop an acute respiratory distress syndrome (ARDS), which requires in the majority of patients a respiratory support with non-invasive mechanical ventilation and, very often, the intubation . Recent evidence is growing in describing the characteristics of this disease, with main focus on lung morphology. Therapeutic strategies implemented for their management may often lead to short-term muscular and functional alterations resulting in ICU-Acquired weakness. These lead to long-term disabilities expressing through dependence and quality of life impairment of survivors. Indeed, few data are still available regarding the peripheral and respiratory muscular characteristics, mainly because this investigation is usually confined in more advance stages of disease. Muscular ultrasonography allows visualization and classification of muscle characteristics which may be described besides muscles' thickness with their echogenicity. In fact, lean muscle tissue has a low echogenicity, whereas intramuscular fat and connective tissue are characterized by a high echogenicity.

Using a greyscale analysis, the total muscle echo-intensity may in fact be quantified. The assumption is that the higher the mean pixel intensity of a muscle region of interest, the lower the muscle quality (i.e., more intramuscular fat or connective tissue) and thus its inhomogeneity. Muscle echogenicity has already been investigated during critical illness, although its modifications over the time and its associated histopathological characteristics remain to be determined. In fact, inflammation and infection as well as fluid shifts may substantially contribute to the increment in muscular inhomogeneity. Few data are available regarding the characteristics of respiratory muscle ultrasound quality during critical illness, as most of the study restricted this methodology to the analysis of peripheral muscles in the detection of ICU acquired weakness. Recently, the parasternal intercostal muscles and the diaphragm have been investigated together in the critical care setting as they represent the easiest accessible respiratory muscles to be investigated by ultrasound .

The investigators hypothesized that a combined assessment of respiratory (i.e., intercostal and diaphragm) and peripheral (i.e., quadriceps) muscles quantity (as measured by thickness) and quality (as assessed by greyscale analysis), would reflect the severity of illness. Thus,the aims of this study are to assess if the quality characteristics of parasternal intercostal, diaphragm and quadriceps muscles of ICU COVID19 patients influenced the outcomes and are correlated with other variables, such as fluid or protein balance, or indexes of inflammation

ELIGIBILITY:
Inclusion Criteria:

- intubated patients with confirmed infection by SARS COV 2 and diagnosis of ARDS

Exclusion Criteria:

* age less than 18 years, history of severe chronic obstructive pulmonary disease, pregnancy, failure to perform respiratory muscle ultrasound

Age Groups: Child, Adult, Older Adult
Study Population: Ards covid19 icu patients
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-02-21 (Actual); Study Completion 2021-02-21 (Actual)

PRIMARY OUTCOMES:
Grayscale and mortality | One year
  assess if the muscular grayscale of parasternal intercostal, diaphragm and quadriceps muscles of ICU COVID19 patients influenced the outcomes

SECONDARY OUTCOMES:
Grayscale and inflammation | One year
  assess if the muscular grayscale characteristics of parasternal intercostal, diaphragm and quadriceps muscles of ICU COVID19 patients are correlated with other variables, such as fluid or protein balance, or indexes of inflammation

CONTACTS AND LOCATIONS:
Locations (1):
- ASST-Santi Paolo e Carlo, San Paolo Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No